CLINICAL TRIAL: NCT04320836
Title: Prospective Study to Determine Evaluate the Validity and Predictive Ability of Physical Exam Signs for Cervical Radiculopathy to Predict Epidural Steroid Injection (ESI) Treatment Outcomes.
Brief Title: Non-organic Signs to Predict Outcomes for Neck Pain
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Washington DC VA Medical Center (Unknown); Seoul National University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00243203
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Cervical Radiculopathy; Cervical Radicular Pain
Keywords: Cervicalgia; Neck pain; Cervical radiculopathy; Cervical radicular pain; Epidural steroid injection; Non-organic sign
MeSH Terms: conditions — Radiculopathy; Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervical epidural steroid injection: This group will receive an interlaminar cervical ESI at C6-7 or C7-T1 with 1 mL steroid (depo-methylprednisolone 40 mg at Johns Hopkins and the DC VA Hospital or dexamethasone 10 mg at Seoul National University) and 2 mL normal saline.
  Interventions: Procedure: Cervical epidural steroid injection

INTERVENTIONS:
Procedure: Cervical epidural steroid injection — Interlaminar cervical epidural steroid injection with steroid and normal saline at C6-7 and C7-T1 (standard of care).

SUMMARY:
Neck pain is the 4th leading cause of disability in the world, with approximately 50% being neuropathic in nature. Epidural steroid injections (ESI) are one of the most commonly used treatments for cervical radiculopathy. Physical exam signs, including non-organic signs, have been shown to predict outcomes for low back pain treatments, but have yet to be adequately studied for neck pain.

In this prospective, observational study, 72 patients with cervical radiculopathy undergoing an initial ESI for this pain episode will undergo a comprehensive history and physical examination that includes the presence of Spurling test, midline and paraspinal tenderness, 9 non-organic tests in 5 categories, and 3 questionnaires to assess depression, anxiety, sleep, and somatization. The investigators will also evaluate patients' MRI results to determine patients' precise pathology. Patients will then receive interlaminar cervical ESI. The primary outcome measure will be the difference in the proportion of people with a positive categorical outcome, defined as a >/= 2-point decrease in arm pain 4 weeks post-procedure coupled with a score >/= 5 on a 7-point patient global impression of change (PGIC) scale 4 weeks post-treatment, indicating subjective improvement.

The main objectives of this study are to:

1. Determine the ability of physical exam, including non-organic signs, to predict ESI outcomes in individuals with cervical radicular pain.
2. Determine the prevalence of different non-organic signs, and the association with other factors that may be associated with non-organic illness such as psychopathology and multiple unrelated pain conditions.

DETAILED DESCRIPTION:
Seventy-two patients with cervical radiculopathy undergoing an initial ESI for this pain episode will undergo a comprehensive history and physical examination that includes the presence of Spurling test, midline and paraspinal tenderness, 9 non-organic tests in 5 categories, and 3 questionnaires to assess depression, anxiety, sleep, and somatization.

Non-organic signs that the investigators will evaluate are:

1. Tenderness

   1. Superficial
   2. Non-anatomical (e.g. cervical radicular pain causing tenderness in the arm or mid-back)
2. Sham stimulation

   1. Downward pressure on head elicits neck pain
   2. With hands clasped behind neck, passive rotation of shoulders elicits neck pain
3. Distraction

   a. Inability to rotate head > 45 degrees during overt range-of-motion testing, but significantly greater range of motion when patient is lying prone and asked to turn head to respond to physician request (e.g. sign paper, count fingers, answer question).
4. Regional disturbances

   1. Sensory disturbances that deviate from normal neuroanatomy or pathology (e.g. single herniated disc causing pain throughout entire arm or radiating into lower back)
   2. Motor disturbances that deviate from normal neuroanatomy or pathology (e.g. dramatic non-neurological weakness, give-away weakness)
5. Overreaction

   1. Verbal (e.g. crying, screaming)
   2. Non-verbal (e.g. exaggerated grimacing, clutching affected area, abnormally slow or rigid movements)

The investigators will evaluate MRI results to determine the precise pathology. Patients will then receive interlaminar cervical ESI. In accordance with standard practice, a Tuohy needle will be directed towards the side of the radicular pain, with correct needle position in the epidural space being confirmed with real-time contrast injection. Once the physician is satisfied with the spread, a 3 mL solution consisting of depo-methylprednisolone 40 mg + 2 mL normal saline will be injected. At Seoul National University, due to Korean healthcare regulations, the mixture will be a 3 mL solution containing 10 mg of dexamethasone and 2 mL saline. The primary outcome measure will be the difference in the proportion of people with a positive categorical outcome, defined as a >/= 2-point decrease in average arm pain 4 weeks post-procedure coupled with a score >/= 5 on a 7-point patient global impression of change (PGIC) scale 4 weeks post-treatment, indicating subjective improvement. Secondary outcome measures will include mean reductions in average and worst 0-10 numerical rating scale (NRS) arm pain scores over the past 7 days, mean reduction in average and worst neck pain scores, neck disability index (NDI) score, medication usage, patient global impression of change (PGIC), Hospital Anxiety and Depression Scale (HADS), Athens Insomnia Scale (AIS), Somatic Symptom Scale-8 (SSS-8), and side effects. Individuals who experience a positive categorical outcome at 4 weeks will continue to be evaluated at 12 weeks, while those with a negative outcome will exit the study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Cervical radicular pain based on history and physical exam (e.g. pain radiating into one or both extremities, sensory loss, muscle weakness, Spurling's test etc.)
* Pain duration > 6 weeks
* Average NRS arm pain score > 4
* MRI evidence of disc pathology consistent with symptoms

Exclusion Criteria:

* Untreated coagulopathy
* Previous spine surgery
* No MRI study
* Epidural steroid injection within past 3 years
* Radiculopathy resulting from tumor or herpes zoster
* Signs or symptoms or myelopathy or spinal cord compression
* Allergic reactions to contrast allergy including macrocyclic gadolinium or depo-methylprednisolone
* Referrals from surgery for diagnostic injections for surgical evaluation
* Serious medical (e.g. congestive heart failure) condition that might preclude optimal outcome
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with clinical and MRI evidence of cervical radicular pain who are scheduled to undergo cervical epidural steroid injection
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Categorical response | 4 weeks
  Positive response is defined as a >/= 2-point reduction in average arm pain coupled with >/= 5/7 score on patient global impression of change. Anything else is a negative response.

SECONDARY OUTCOMES:
Average arm pain | 4 weeks
  Average arm pain on 0-10 numerical rating scale.
Worst arm pain | 4 weeks
  Worst arm pain on 0-10 numerical rating scale.
Average neck pain | 4 weeks
  Average neck pain on 0-10 numerical rating scale.
Worst neck pain | 4 weeks
  Worst neck pain on 0-10 numerical rating scale.
Neck disability index (NDI) score | 4 weeks
  NDI Score on 0-10 numerical rating scale.
Somatic Symptom Scale (SS-8) score | 4 weeks
  8-question survey, out of 32 points measuring somatization.
Athens Insomnia Scale (AIS) score | 4 weeks
  8-question survey, out of 24 points measuring sleep quality.
Hospital Anxiety and Depression Scale (HADS) | 4 weeks
  14-question survey measuring anxiety and depression (each out of 21 points).
Patient Global Impression of Change (PGIC) scale | 4 weeks
  7-point Likert scale measuring patient-reported improvement.
Patient Global Impression of Change (PGIC) scale | 12 weeks
  7-point Likert scale measuring patient-reported improvement.
Hospital Anxiety and Depression Scale (HADS) | 12 weeks
  14-question survey measuring anxiety and depression (each out of 21 points).
Athens Insomnia Scale (AIS) score | 12 weeks
  8-question survey, out of 24 points measuring sleep quality.
Somatic Symptom Scale (SS-8) score | 12 weeks
  8-question survey, out of 32 points measuring somatization.
Average arm pain | 12 weeks
  Average arm pain on 0-10 numerical rating scale.
Worst arm pain | 12 weeks
  Worst arm pain on 0-10 numerical rating scale.
Average neck pain | 12 weeks
  Average neck pain on 0-10 numerical rating scale.
Worst neck pain | 12 weeks
  Worst neck pain on 0-10 numerical rating scale.
Neck disability index (NDI) score | 12 weeks
  NDI Score on 0-10 numerical rating scale.
Categorical response | 12 weeks
  Positive response is a >/= 2-point reduction in average arm pain coupled with >/= 5/7 score on patient. Anything else is a negative response.

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Cohen, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (2):
  - DC VA Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins, Baltimore, Maryland
- Seoul National University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Upon request
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Up to 3 years after publication
Access Criteria: Upon request, contingent on objectives

REFERENCES:
- [Background] Fishbain DA, Cole B, Cutler RB, Lewis J, Rosomoff HL, Rosomoff RS. A structured evidence-based review on the meaning of nonorganic physical signs: Waddell signs. Pain Med. 2003 Jun;4(2):141-81. doi: 10.1046/j.1526-4637.2003.03015.x. PMID 12911018
- [Background] Waddell G, McCulloch JA, Kummel E, Venner RM. Nonorganic physical signs in low-back pain. Spine (Phila Pa 1976). 1980 Mar-Apr;5(2):117-25. doi: 10.1097/00007632-198003000-00005. PMID 6446157
- [Background] Jorritsma W, Dijkstra PU, De Vries GE, Geertzen JH, Reneman MF. Physical dysfunction and nonorganic signs in patients with chronic neck pain: exploratory study into interobserver reliability and construct validity. J Orthop Sports Phys Ther. 2014 May;44(5):366-76. doi: 10.2519/jospt.2014.4715. Epub 2014 Apr 14. PMID 24730436
- [Derived] Cohen SP, Doshi TL, Dolomisiewicz E, Reece DE, Zhao Z, Anderson-White M, Kasuke A, Wang EJ, Hsu A, Davis SA, Yoo Y, Pasquina PF, Moon JY. Nonorganic (Behavioral) Signs and Their Association With Epidural Corticosteroid Injection Treatment Outcomes and Psychiatric Comorbidity in Cervical Radiculopathy: A Multicenter Study. Mayo Clin Proc. 2023 Jun;98(6):868-882. doi: 10.1016/j.mayocp.2022.11.022. Epub 2023 Feb 15. PMID 36803892